CLINICAL TRIAL: NCT05497817
Title: Fostering Caregiver Connections Via Intentional Technology Pairing for Caregivers of Patients With Alzheimer's Disease and Other Types of Dementia-Phase 2
Brief Title: A Study to Evaluate Caregiver Connections Via Technology for Patients With Alzheimer's and Other Types of Dementia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn and being modified under another protocol
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Minnesota HealthSolutions (Industry)
Responsible Party: Principal Investigator, Julie A. Fields, Ph.D., L.P., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20-013202; R44AG065088 (NIH)
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Caregiver Stress; Dementia; Alzheimer Dementia; Lewy Body Dementia; Parkinson Disease Dementia; Frontotemporal Dementia
MeSH Terms: conditions — Caregiver Burden; Dementia; Alzheimer Disease; Lewy Body Disease; Frontotemporal Dementia | interventions — Algorithms

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to two different arms of the study: one where the algorithm matches individuals and one where matches are randomly assigned.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Algorithmically Matched (Experimental): Individuals that identify as a current and/or former Care Partner for a person with dementia will be matched to other care partners using an algorithm based on personal preferences.
  Interventions: Behavioral: Algorithm
- Randomly Matched (Active Comparator): Individuals that identify as a current and/or former Care Partner for a person with dementia will be randomly matched to other care partners.
  Interventions: Behavioral: Random Match

INTERVENTIONS:
Behavioral: Algorithm — Current and/or former Care Partners of persons with dementia will be matched using an algorithm to other Care Partners who might provide emotional support.
  Arms: Algorithmically Matched
Behavioral: Random Match — Current and/or former Care Partners of persons with dementia will be randomly matched to other Care Partners who might provide emotional support.
  Arms: Randomly Matched

SUMMARY:
This research is being done to develop a unique matching process for caregivers of persons living with dementia, such as Alzheimer's disease, Lewy body dementia, frontotemporal degeneration, or other dementia syndromes. Dementia caregivers often assume greater caregiving burden than do non-dementia caregivers, and the caregiving duration tends to be longer. Many caregivers do not have the adequate support they need. Peer-to-peer support has been shown to improve quality of life, increase use of services, improve caregiver health, and reduce hospitalizations in the person they are caring for. This study will assess a technology platform and matching process for the purpose of peer-to-peer emotional support aimed at improving overall wellbeing in dementia care partners/caregivers.

ELIGIBILITY:
Individuals in a current or former caregiving role for a family member living with dementia will be recruited for this study. There will be no sex or gender restrictions, or exclusion based on race or ethnicity. Participants must be at least 18 years of age.

Inclusion Criteria:

* The participant must have a family member that has been diagnosed with dementia.
* The participant must identify as a Care Partner or Caregiver who has contact with their loved one with dementia, in person or by phone, and who provides social/emotional support and full or partial assistance with daily activities at least 3 days per week.
* The participant must have been caring for their loved one with dementia for at least 3 months.
* All participants must have access to a computer and be able to use the internet.
* All participants must be English speaking.
* All participants must agree to participate in the 15-month study, which includes completing questionnaires, brief "virtual" interactions with the study coordinator quarterly, and actively interacting with the website and potential matches.
* All participants must agree to follow-up contact throughout the duration of the study, which is anticipated to last 3 years.

Exclusion Criteria:

* Care Partner's loved one does not have a confirmed diagnosis of dementia.
* Care Partner is unable to provide consent.
* Care Partner was or has been in that role for less than 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Match Satisfaction Questionnaire | 12 months
  All participants will complete a match satisfaction questionnaire to assess whether being matched to a supportive Care Partner via an algorithm based on personal preferences results in greater match satisfaction than being matched at random.
Change over time from Baseline Resilience to 12 months | Baseline,12 months
  All participants will complete questions surveying resilience to determine whether Care Partners randomized to algorithmic matching based on personal preferences will report a greater sense of resiliency after being matched than Care Partners who are randomly matched.
Change over time from Baseline Quality of Life to 12 months | Baseline, 12 months
  All participants will complete questions surveying quality of life to determine whether Care Partners randomized to algorithmic matching based on personal preferences will report improved quality of life after being matched than Care Partners who are randomly matched.
Scale of Perceived Social Support | 12 months
  All participants will complete survey questions regarding perceived level of social support to assess impact on match satisfaction.

SECONDARY OUTCOMES:
Survey of Executive Skills | 12 months
  All participants will complete questions regarding executive functioning (e.g., flexibility, problem-solving) to determine whether the level of these skills relates to ease or difficulty in finding a satisfactory supportive Care Partner match.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Fields, PhD, LP, Principal Investigator — Mayo Clinic; Kevin Kramer, PhD, Principal Investigator — Minnesota HealthSolutions, Inc.

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials